CLINICAL TRIAL: NCT03097744
Title: Predictors of Early Success From Circumferential Compression STITCH Meniscal Repairs
Acronym: STITCHRetro
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CTX-CP003
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2019-01

CONDITIONS: Knee Medial Meniscus Tears; Meniscus Lesion; Meniscus; Rupture, Bucket Handle; Meniscus Disorder
Keywords: Lateral Meniscus Tear; Medial Meniscus Tear
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Ceterix NovoStitch — The device allows the physician to place a circumferential compression stitch around meniscal tears. This stitch is placed by passing suture from the tibial side to the femoral side of the meniscus and across the tear. This allows compression across the entire tear surface.

SUMMARY:
This is a retrospective study of meniscal tear repairs at least one-year post repair status. All patients were treated with Ceterix NovoStitch devices. The primary objectives of this study are to assess the clinical repair success rate via reoperation and PROs at greater than 12 months.

DETAILED DESCRIPTION:
The study is a retrospective, non-randomized, single-group assignment, open-label study of repairs of meniscal tears status post repair. The following clinical efficacy endpoints will be evaluated at greater than 12 months:

* Reoperation rate
* Validated patient-reported outcomes measures
* Contribution of the following retrospective covariates on failure and outcomes when available: Type of tear, Location of tear (lateral versus medial), Chronicity of symptoms, Nature of tear (degenerative versus traumatic), Length of tear, Patient age, Patient gender, Length of rehabilitation protocol, Performance of trephination, Inclusion of biologic enhancement, Meniscal repair alone versus meniscal repair combined with ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give consent by voluntarily providing written informed consent in accordance with governing Institutional Review Board (IRB)/Independent Ethics Committee (IEC) requirements, local regulations, and Health Insurance Portability and Accountability Act (HIPAA) Authorization (or equivalent if locally applicable)
* In the opinion of the Investigator are able to comply with study-required follow-up

Exclusion Criteria:

* Post-operative interval <1year
* Concurrent bony fractures
* Post-operative reinjury (except the meniscus)
* Pre-operative arthritis grade 3 or higher on modified outerbridge
* Knee surgery prior to meniscus repair surgery
* Any kind of infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals, 18-years-old or older, who have undergone a meniscus repair with a Ceterix NovoStitch device at least 12 months ago.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Reoperation Rate | January 2015-February 2016
  Data provided by patients
Validated patient-reported outcomes measures | January 2015-February 2016
  IKDC Subjective
Contribution of the following retrospective covariates on failure and outcomes when available | January 2015-February 2016
  Type of tear Location of tear (lateral versus medial), Chronicity of symptoms, Nature of tear (degenerative versus traumatic), Length of tear, Patient age, Patient gender, Length of rehabilitation protocol, Performance of trephination, Inclusion of biologic enhancement, Meniscal repair alone versus meniscal repair combined with ACL reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Olson, Study Director — Ceterix Orthopaedics
Locations (1):
- Agility Center Orthopedics, Bentonville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saliman JD. The circumferential compression stitch for meniscus repair. Arthrosc Tech. 2013 Jul 12;2(3):e257-64. doi: 10.1016/j.eats.2013.02.016. eCollection 2013. PMID 24265995
- [Background] Nepple JJ, Dunn WR, Wright RW. Meniscal repair outcomes at greater than five years: a systematic literature review and meta-analysis. J Bone Joint Surg Am. 2012 Dec 19;94(24):2222-7. doi: 10.2106/JBJS.K.01584. PMID 23318612